CLINICAL TRIAL: NCT00043615
Title: Acquisition of Blood, Bone Marrow, Tumor, or Tissue Samples
Brief Title: Collection of Blood, Bone Marrow, Tumor or Tissue Samples
Status: Completed | Type: Observational
Sponsor: National Cancer Institute (NCI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 020258; 02-C-0258; NCT00896805 (obsolete NCT alias)
Record Dates: First submitted 2002-08-09; First posted 2002-08-12 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2012-04-10

CONDITIONS: Neoplasms; Precancerous Conditions
Keywords: Angiogenesis; Drug Resistance; Signal Transduction; EGFR; Survival Factors; Malignancy; Pre-Cancer Condition; Cancer Risk
MeSH Terms: conditions — Neoplasms; Precancerous Conditions

SUMMARY:
This study will collect biological samples-blood, bone marrow, tumor or other tissue samples-for use in cancer-related research. The specimens will be used for various tests of drug resistance, blood vessel formation, cancer-causing proteins and immune functions. The purpose is to identify steps in the cancer development process that may serve as targets for treatment and to test various therapies for current and future cancer treatment clinical trials.

Individuals 18 years of age and older with cancer or a pre-cancerous condition, such as colon polyps or cervical dysplasia, are eligible for this study, as are patients at high risk for cancer. In addition, patients who do not have cancer but require surgery, biopsy or other procedure for another medical reason may be included as normal specimen donors.

Participants will have about 40 milliliters (3 tablespoons) of blood drawn upon entering the study and additional 40-ml samples drawn periodically during the course of treatment. No more than 120 ml of blood will be drawn over a 12-month period. Some patients may require a surgical procedure or biopsy (removal of tumor tissue) for medical reasons or as part of their enrollment in a research treatment study. In such cases, a portion of the specimens collected during those procedures will be used for the research studies in this protocol.

DETAILED DESCRIPTION:
Patients will be evaluated at NNMC Clinics. Blood samples may be collected at the initial visit and at follow-up visits. Tumor samples may be obtained by fine needle aspirate, by removal of pleural or peritoneal fluid, or by excisional biopsy, or other procedure. In general, biopsy tissue will be obtained as an additional sample at the time of a medically indicated procedure. In some cases, a biopsy may be performed only to obtain a research sample providing the tumor is accessible with a minimal risk to the patient. Specific risks will be described in a separate consent to be obtained at the time of the biopsy. Tumor samples and blood samples will be processed and/or stored for use in research efforts in the laboratories of the Medical Oncology Branch, Experimental Transplant and Immunology Branch, or Genetics Branch, Center for Cancer Research, NCI at Navy and NIH.

ELIGIBILITY:
* INCLUSION CRITERIA:

Patients must have a performance status of ECOG greater than or equal to 3 for admission to this protocol.

Subjects must be at least 18 years old.

Patients with any malignancy, high-risk, pre-malignant condition (for example, colonic polyps, cervical dysplasia, atypical ductal hyperplasia or oral leukoplakia), undergoing reduction mammoplasty or prophylactic mastectomy are eligible.

Patients requiring a surgical procedure for any medical indication can be included on study. These patients would be considered normal donors (no diagnosis of cancer).

Patients requiring biopsy or any procedure for any medical indication can be included on study. These patients will be considered normal donors (no diagnosis of cancer).

Patients not requiring biopsy for a medical indication can be included on the study solely for the purpose of obtaining research samples, including blood, pleural fluid, or peritoneal fluid, or biopsy samples, providing the biopsy or aspiration procedure is of minimal risk, i.e., fine needle aspirate, bone marrow aspirate, or excisional biopsy.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 74 (Actual)
Dates: Start 2002-07-29; Study Completion 2012-04-10

CONTACTS AND LOCATIONS:
Overall Officials: Kevin A Camphausen, M.D., Principal Investigator — National Cancer Institute (NCI)
Locations (2):
- United States (2):
  - National Naval Medical Center, Bethesda, Maryland
  - National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland